CLINICAL TRIAL: NCT06716060
Title: Prevalence of Intestinal Parasitic Infections in Under-Five Children With Malnutrition in Sohag, Egypt
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Mahmoud, Prevalence of Intestinal Parasitic Infections in Under-Five Children with Malnutrition in Sohag, Egypt, Sohag University
Other Study IDs: Soh-Med-24-08-MS
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Malnutrition, Child
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to estimate the prevalence of intestinal parasitic infections in under-five children with malnutrition.

DETAILED DESCRIPTION:
Malnourished children are vulnerable to IPIs suffering. In contrast, IPIs can contribute considerably to the evolution of undernutrition in the pediatric population, thus creating a potentially lethal cycle/vicious cycle of worsening illness and deteriorating nutritional status so, I will examine stool specimens of those children suffering from malnutrition.

One fecal sample will be collected from each patient in a labelled clean plastic container. Specimens will be immediately transferred to the Medical Parasitology Department laboratory The obtained fecal samples will be both macroscopically and microscopically examined. For microscopic examination, specimens will be examined by direct smear and FECT.

Anthropometric indices will be used for checking the nutritional status of the recruited children.

ELIGIBILITY:
Inclusion Criteria:

- 100 children aged between 6 months and 5 years, having malnutrition symptoms (growth retardation, failure to thrive, lethargy, generalized weakness, xerophthalmia, etc.) will be randomly recruited from pediatric outpatient clinics, Faculty of medicine, Sohag University.

Exclusion Criteria:

* children who took specific anthelmintic, antiprotozoal, purgatives or anti-diarrheal drugs three weeks before the stool sampling.

Ages: 6 Months to 5 Years | Sex: All
Age Groups: Child
Study Population: - 100 children aged between 6 months and 5 years, having malnutrition symptoms (growth retardation, failure to thrive, lethargy, generalized weakness, xerophthalmia, etc.)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Intestinal Parasitic Infections in Under-Five Children with Malnutrition in Sohag, Egypt | 10 months
  Malnourished children are vulnerable to IPIs suffering. In contrast, IPIs can contribute considerably to the evolution of undernutrition in the pediatric population, thus creating a potentially lethal cycle/vicious cycle of worsening illness and deteriorating nutritional status so, I will examine stool specimens of those children suffering from malnutrition.
  Malnourished children are vulnerable to IPIs suffering. In contrast, IPIs can contribute considerably to the evolution of undernutrition in the pediatric population, thus creating a potentially lethal cycle/vicious cycle of worsening illness and deteriorating nutritional status so, I will examine stool specimens of those children suffering from malnutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Esraa Ahmed Mahmoud Mohamed, Sohag, Saqulta, Egypt